CLINICAL TRIAL: NCT03577327
Title: The Gut and Skin Microbiome in Vitiligo Disease Progression
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, I Caroline Le Poole, Professor, Northwestern University
Other Study IDs: ICLP10302017
Record Dates: First submitted 2018-04-02; First posted 2018-07-05 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Vitiligo; Healthy
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adults with vitiligo
- Healthy adults

SUMMARY:
Investigators plan to perform a pilot study that aims to characterize the microbiome of human vitiligo patients with both active and stable disease and compare this to the microbiome of age and sex matched controls. The investigators aim to answer the question whether the gut and skin microbiome of patients with vitiligo differs from the general population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with and/or without vitiligo lesional expansion over the past year.
* Age/sex-matched controls who do not have a diagnosis of vitiligo
* Subjects who are age 18-89 years of age at time of enrollment
* Subjects who are able and willing to give informed consent for this study and the Dermatology Tissue Acquisition and Biorepository (STU00009443)

Exclusion Criteria:

* Subjects who are younger than 18 years of age or 90 years of age or older
* Subjects who are unable to give consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with or without vitiligo who are under the age of 90 years old.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Microbiome composition | 12 months
  Diversity analysis of microbiome samples in control subjects versus vitiligo subjects (measured by number of bacteria species/sample)
Disease Progression | 12 months
  Disease progression in control subjects versus vitiligo subjects (measured by VASI score (0-100)).

SECONDARY OUTCOMES:
Diet History Food Frequencies | 12 months
  Scoring from diet history food frequency questionnaires (measured by average daily food frequency scores).

CONTACTS AND LOCATIONS:
Overall Officials: I. Caroline Le Poole, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No